CLINICAL TRIAL: NCT06288100
Title: The Effect of Open Wedge High Tibial Osteotomy on the Posterior Tibial Slope In Skeletally Mature Patient
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelfattah Abbas, Mohamed Abdelfattah Abbas, Al-Azhar University
Other Study IDs: OWHTOPTS
Record Dates: First submitted 2024-02-15; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Genu Varum
MeSH Terms: conditions — Genu Varum | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observations: number of patients, sex, age, Bodi Mass Index , Range of Motion ,type of plate & Screws used , Degree of deformity .
  Digital radiography (General Electric Healthcare ) functional scores software T-tests, One-way analysis of variance.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — 1. Measure changes in tibial slope after medial opening wedge High tibial osteotomy in Skeletally mature patient with unicompartmental osteoarthitis and genuvarus knee
  2. Evaluate the effect of tibial slope angle change on the clinical outcome at 1 year .

SUMMARY:
High tibial osteotomy has been established as an efficient surgical intervention for young patients with uni-compartmental osteoarthritis of the knee. The principle of this surgery involves the realignment of the lower extremity to shift the load distribution from the medial compartment into the lateral compartment, thus leading to a decrease in symptoms related to medial compartment knee Osteoarthritis However, medial opening wedge high tibial osteotomy is also known to affect the posterior tibial slope angle , and it is reported that posterior tibial slope angle increases after medial opening wedge high tibial osteotomy .

DETAILED DESCRIPTION:
High tibial osteotomy has been established as an efficient surgical intervention for young patients with uni-compartmental osteoarthritis of the knee. Medial opening wedge high tibial osteotomy is a well established surgery for patients with medial compartment knee osteoarthritis its most notable advantages include the precision of intraoperative angular correction, absence of the risk of peroneal nerve palsy in fibular osteotomy, absence of leg shortening, and preservation of bone stock.

The principle of this surgery involves the realignment of the lower extremity to shift the load distribution from the medial compartment into the lateral compartment, thus leading to a decrease in symptoms related to medial compartment knee Osteoarthritis However, medial opening wedge high tibial osteotomy is also known to affect the posterior tibial slope angle , and it is reported that posterior tibial slope angle increases after medial opening wedge high tibial osteotomy .

Satisfactory outcomes after surgery require optimal realignment both in the sagittal and coronal planes; in fact, poor realignment could lead to unsatisfactory clinical outcomes. An unintentional increase in posterior tibial slope angle after medial opening wedge high tibial osteotomy may influence knee kinematics and stability in the sagittal plane, which could lead to anterior translation of the tibial plateau, anterior shift of the tibiofemoral contact area, and subsequent redistribution of pressure into the posterior tibial plateau (particularly in knees with injured anterior cruciate ligaments). These conditions could result in articular cartilage degradation and further knee disability

ELIGIBILITY:
Inclusion criteria

* Age: 20 : 65 years
* Genuvarus deformity
* 70° of range of motion
* Medial uni-compartmental osteoarthritis.

Exclusion criteria

* Posterior instability (relating to the posterior cruciate ligament)
* Body Mass Index under 30
* Sever Genuvarus > 20 degree

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data Collection:
  The study and patients were collected according to number of patients, sex, age, Bodi Mass Index , Range of Motion ,type of plate & Screws used , Degree of deformity . Digital radiography, functional scores, software was used for statistical analysis. compare the Posterior Tibial Slope between the different Posterior Tibial Slope sides and sexes. One-way analysis of variance was used to compare the Posterior Tibial Slope between the different age groups. Posterior Tibial Slope was evaluated in all studies according to radiographic.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
The Effect of Open Wedge High Tibial Osteotomy on the Posterior Tibial Slope In Skeletally Mature Patient | Measure Posterior tibial slope by X Ray in Lateral View and Evaluate the effect of tibial slope angle change on the clinical outcome at 1 year
  Measure changes in tibial slope after medial opening wedge High tibial osteotomy in Skeletally mature patient with unicompartmental osteoarthitis and genuvarus knee Evaluate the effect of tibial slope angle change on the clinical outcome at 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Abdelfattah Abbas, Asyut, Egypt